CLINICAL TRIAL: NCT06989151
Title: A Pilot Study of Cognitive Remediation Therapy for Autistic Adolescents
Brief Title: Cognitive Remediation for Autistic Adolescents
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 338473
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Single arm for pilot study
  Interventions: Behavioral: Cognitive Remediation Therapy

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — 8 session psychological intervention.

SUMMARY:
Autistic youth have extremely high levels of co-occurring mental health difficulties, including rates of depression and anxiety which are between two and four times more common compered to non-autistic people. Cognitive inflexibility is a characteristic which is strongly associated with higher levels of anxiety and depression in autism. Currently, there are no existing treatments which can promote flexible thinking. Cognitive Remediation Therapy is a promising intervention which has been used with different patient groups to improve flexibility. This study aims to develop and adapt the current CRT treatment for use with autistic youth and then conduct a pilot study with 20 participants.

DETAILED DESCRIPTION:
The existing evidence that CRT is effective for those with autistic features leads us to hypothesize that with minor adaptations the intervention will be acceptable to those with autism. Given the strong association between CI and anxiety (and other internalizing difficulties such as depression; ref) by targeting this specific trait it is hypothesized that an adapted CRT will a) increase flexible thinking and b) reduce symptoms of anxiety and depression.

Key objectives:

1. To use the existing literature of adapted interventions for autism and input from autistic youth and their parents to adapt CRT for use with autistic youth.
2. To establish the acceptability of adapted CRT by conducting a proof-of-principle pilot study.
3. To gather preliminary outcome data on CI, anxiety and depression, and other key measures such as levels of functional outcomes to inform the design of an acceptability and feasibility RCT for future funding applications.

Methods:

Participants will all complete 8 adapted CRT intervention sessions held twice weekly. Outcome measures will be collected pre- and post intervention. Measures of acceptability of the intervention (e.g., retention rate) will be recorded and qualitative interviews will gather feedback on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 12-16 years of age with a confirmed clinical diagnosis of autism (based on verified diagnostic report).
* Verbal/intellectual ability in average range
* Sufficient spoken English to access the intervention.
* Young person must be under the care of a local mental health service who can respond to any changes in routine clinical care / risk issues that arise.

Exclusion Criteria:

* Not currently receiving alternative psychological intervention
* Not actively self-harming or deemed at risk to themselves or others

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Acceptability 1 - Drop out rate | 8 weeks
  Number of participants who drop-out from the study
Acceptability 2 - session attendance rate: | 8 weeks
  total number of sessions attended out of a maximum of 8 per participant
Acceptability 3 - adherence to the therapy protocol | 8 weeks
  Completion rates of between session work - recorded as percentage.
Acceptability 4 - Semi-structured qualitative interviews post intervention | 8 weeks

SECONDARY OUTCOMES:
Cognitive Flexibility Scale | 8 weeks
  Questionnaire measure of flexibility
DFLEX | 8 weeks
  Detail and Flexibility Questionnaire
Revised Child Anxiety and Depression Scale | 8 weeks
Mood and Feelings Questionnaire | 8 weeks
Work and Social Adjustment Scale | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No